CLINICAL TRIAL: NCT03252184
Title: Effects of Photobiomodulation on Endothelial Function, Blood and Endothelial Markers, and Nitric Oxide Metabolites in Healthy Subjects.
Brief Title: Effects of Photobiomodulation on Endothelial Function in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rodrigo Della Méa Plentz (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Della Méa Plentz, Principal Investigator, Federal University of Health Science of Porto Alegre
Organization: Federal University of Health Science of Porto Alegre (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBMLLLT
Record Dates: First submitted 2017-05-18; First posted 2017-08-17 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Healthy Behavior
Keywords: Phototherapy; Laser Therapy; Endothelium-Dependent; Vascular Endothelium; Low Intensity Light Therapy; Relaxing Factors
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The study will be separated in phases in according to photobiomodulation device employed. Initially, we will use the laser with 658nm, power output of 10mW per point and fluence of 18J, 36J e 54J per area. The individuals will be randomly assigned to: group 1 (energy dose of 18J), group 2 (energy dose of 36J), group 3 (energy dose of 54J), and group 4 (placebo). In the second phase, we will use the laser with 810nm, power density of 714 mW/cm2 and fluence of 30 J per spot. The individuals will be randomly assigned to: group 1 (energy dose of 30J), group 2 (energy dose of 60J) and group 3 (placebo). Finally, we will measure the time of blood vessel dilation after photobiomodulation with 30J and 60J.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Phase 1 - Low level laser therapy - 1 (G1) (Experimental): Low level laser therapy with energy dose of 18J will be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 1
- Phase 1 - Low level laser therapy - 1 (G2) (Experimental): Low level laser therapy with energy dose of 36J will be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 1
- Phase 1 - Low level laser therapy - 1 (G3) (Experimental): Low level laser therapy with energy dose of 54J will be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 1
- Phase 1 - Placebo low level laser therapy - 1 (G4) (Placebo Comparator): Low level laser therapy with equipment turn off (placebo) be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 1
- Phase 2 - Low level laser therapy - 2 (G1) (Experimental): Low level laser therapy with energy dose of 30J will be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 2
- Phase 2 - Low level laser therapy - 2 (G2) (Experimental): Low level laser therapy with energy dose of 60J will be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 2
- Phase 2 - Placebo low level laser therapy - 2 (G3) (Placebo Comparator): Low level laser therapy with equipment turn off (placebo) be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 2
- Phase 3 - Low level laser therapy - 3 (G1) (Experimental): Low level laser therapy with energy dose of 30J will be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 3
- Phase 3 - Low level laser therapy - 3(G2) (Experimental): Low level laser therapy with energy dose of 60J will be applied on left brachial artery of the subject.
  Interventions: Device: Low level laser therapy - 3

INTERVENTIONS:
Device: Low level laser therapy - 1 — In the phase 1, the low level laser therapy will be performed with the Fluence device (HTM, Brasil) and the probe from the same manufacturer. For the interventions in groups G1, G2 and G3 (photobiomodulation) will be used, respectively, the energy doses of 18J, 36J and 54J. A 658nm wavelength with an output power of 10mW will be used. Group 4 intervention (placebo photobiomodulation) will be performed with the application of the device turned off. Each intervention will be performed in one day, with an interval of two days between each intervention. Photobiomodulation will be performed on the region of the radial and ulnar arteries of the left arm of each individual. The laser probe will be placed in direct contact with the skin.
  Other Names: Photobiomodulation; LLLT
  Arms: Phase 1 - Low level laser therapy - 1 (G1); Phase 1 - Low level laser therapy - 1 (G2); Phase 1 - Low level laser therapy - 1 (G3); Phase 1 - Placebo low level laser therapy - 1 (G4)
Device: Low level laser therapy - 2 — In the phase 2, the low level laser therapy will be performed with the Thor DD2 (London, UK) and the cluster probe from the same manufacturer. For the interventions in groups G1 and G2 (photobiomodulation) will be used, respectively, the energy doses of 30J and 60J. A 810nm wavelength and an output power of 200mW will be used. Group 3 intervention (placebo photobiomodulation) will be performed with the application of the device turned off. Each intervention will be performed in one day, with an interval of two days between each intervention. Photobiomodulation will be performed on the region of the radial and ulnar arteries of the left arm of each individual. The laser probe will be placed in direct contact with the skin.
  Other Names: Photobiomodulation; LLLT
  Arms: Phase 2 - Low level laser therapy - 2 (G1); Phase 2 - Low level laser therapy - 2 (G2); Phase 2 - Placebo low level laser therapy - 2 (G3)
Device: Low level laser therapy - 3 — In the phase 3, the low level laser therapy will be performed with the Thor DD2 (London, UK) and the cluster probe from the same manufacturer. For the interventions in groups G1 and G2 (photobiomodulation) will be used, respectively, the energy doses of 30J and 60J. A 810nm wavelength and an output power of 200mW will be used. Each intervention will be performed in one day, with an interval of two days between each intervention. Photobiomodulation will be performed on the region of the radial and ulnar arteries of the left arm of each individual. The laser probe will be placed in direct contact with the skin.
  Other Names: Photobiomodulation; LLLT
  Arms: Phase 3 - Low level laser therapy - 3 (G1); Phase 3 - Low level laser therapy - 3(G2)

SUMMARY:
The endothelial cell layer is responsible for the control of vascular homeostasis, a process mediated by vasoconstricting and vasodilatory substances. The principal endothelium-dependent vascular dilator is nitric oxide (NO), and the reduction of its synthesis or bioavailability is the main cause for the development of endothelial dysfunction. The use of photobiomodulation may be beneficial in several clinical situations. At the endothelial level, the stimulatory effects on vascular endothelial growth factor, NO secretion, number of capillaries and proliferation of endothelial cells are outstanding. The objective of this study is to evaluate the effects of photobiomodulation on the arterial endothelial function of healthy individuals. The study design will be a randomized, crossover, clinical trial and the sample will be composed of subjects selected by the eligibility criteria, and randomly randomized according to the order of intervention of the groups. The hypothesis is that at the end of the protocol with photobiomodulation an increase in endothelial function and blood markers of endothelial function occurs, and no tissue temperature variation.

DETAILED DESCRIPTION:
Detailed Description: The endothelial cell layer is responsible for the control of vascular homeostasis, a process mediated by vasoconstricting and vasodilatory substances. The principal endothelium-dependent vascular dilator is nitric oxide (NO), and the reduction of its synthesis or bioavailability is the main cause for the development of endothelial dysfunction. The use of photobiomodulation may be beneficial in several clinical situations. At the endothelial level, the stimulatory effects on vascular endothelial growth factor, NO secretion, number of capillaries and proliferation of endothelial cells are outstanding. It has also been shown an increase in glutathione levels, antioxidant effect and angiogenic potential, which shows a potential vascular effect, and consequently, an improvement in endothelial function. The objective of this study is to evaluate the effects of photobiomodulation on the arterial endothelial function of healthy individuals. The study design will be a randomized, crossover, clinical trial and the sample will be composed of 16 healthy subjects selected by the eligibility criteria, and randomly randomized according to the order of intervention of the groups. The hypothesis is that at the end of the irradiation protocol with photobiomodulation an increase in endothelial function and blood markers of endothelial function occurs, and no tissue temperature variation. The primary objective is to evaluate the effects of photobiomodulation on the arterial endothelial function of healthy individuals. The secondary objectives are: 1) To evaluate the time of blood vessel dilation after photobiomodulation. 2) To evaluate the effects of photobiomodulation on blood markers (hemogram) and endothelial markers (cGMP and L-arginine), and Nitric oxide (nitrite and nitrate). 3) To analyze associations between markers and metabolites with endothelial function due to the effects of Photobiomodulation. 3) Analyze the local temperature before and after photobiomodulation. 4) Analyze the local temperature before and after the measurement of Endothelial function. 5) Evaluate possible associations between blood and endothelial markers, nitric oxide pathway metabolites and Endothelial function with local temperature. 6) To compare the effects of energy doses and wavelenghts of photobiosmodulation on endothelial function, blood and endothelial markers, and metabolites of the nitric oxide pathway. The research will be developed in room 709 of the Laboratory of Physiotherapy in building II, UFCSPA and, for randomization, the simple technique will be used through numbers generated by a freely available software. The generation of the sequence of numbers will be done by a blind researcher, after the selection of the individuals by the eligibility criteria. The study will be separated in phases in according to photobiomodulation device employed. Initially, we will use the laser with 658nm, power output of 10mW per point and fluence of 18J, 36J e 54J per area. The individuals will be randomly assigned to: group 1 (energy dose of 18J), group 2 (energy dose of 36J), group 3 (energy dose of 54J), and group 4 (placebo). In the second phase, we will use the laser with 810nm, power density of 714 mW/cm2 and fluence of 30 J per spot. The individuals will be randomly assigned to: group 1 (energy dose of 30J), group 2 (energy dose of 60J) and group 3 (placebo). Finally, we will measure the time of blood vessel dilation after photobiomodulation with 30J and 60J. The normality of the data will be evaluated by the Shapiro-Wilk test. Data with symmetrical distribution will be presented as mean ± standard deviation, and data with asymmetric distribution as median and interquartile range (P25 - P75). The baseline characteristics of the patients will be compared by Student's t-test or Mann-Whitney when the distributions are parametric or non-parametric, respectively. The categorical variables will be compared by the Chi-square test. Variance Analysis (ANOVA) will be used for repeated measures for pre and post-intervention data analysis, or the Mann-Whitney test (asymmetric distribution), followed by Bonferroni post hoc. The Pearson or Sperman correlations will be used for possible association between the analyzed variables. Statistical significance of 5% (p <0.05) will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years
* Body mass index (BMI: kg / m2) lower than 30
* Absence of symptoms of musculoskeletal disorders
* No use of medications
* Non-smokers and / or alcoholics
* Absence of previous diagnosis of diseases Rheumatological, cardiovascular, renal, metabolic, neurological, oncological, immunological, hematological, psychiatric or cognitive.

Exclusion Criteria:

On the days of evaluation and intervention:

* Individuals who performed high intensity physical activity in the previous 72 hours
* Individuals who had an inflammatory response (> 3 mg / dL, fibrinogen <200 or> 400mg / dL) or leukocytosis (> 11,000 x103 / Mm3)
* Individuals who have consumed caffeine, juices or citrus fruits, high-fat foods and alcohol in the 12 hours prior to the test
* Individuals who are not fasting for 12 hours
* Individuals who have used anti-inflammatory, antipyretic or analgesic drugs
* Individuals who having an arterial diameter <0.25 mm or> 5.0 mm
* Individuals with present endothelial dysfunction evaluated by the FMD technique (dilation <8%).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in arterial endothelial function | The evaluation of the arterial endothelial function will be performed 20 minutes before and 20 minutes after the intervention with photobiostimulation
  The assessment of arterial endothelial function will be performed through the technique of flow-mediated dilatation, by high resolution ultrasound

SECONDARY OUTCOMES:
Change in body temperature | The evaluation of the arterial endothelial function will be performed 15 minutes before and 15 minutes after the intervention with photobiostimulation
  The local temperature will be evaluated by thermography
Change in inflammatory profile | Basal blood collection (5 minutes before) and immediately after each intervention (5 minutes after)
  The inflammatory profile will be evaluated by C-reactive protein dosage
Change in arterial endothelial function (vasodilatation) | Basal blood collection (5 minutes before) and immediately after each intervention (5 minutes after)
  The vasodilatation will be evaluated by nitrite/nitrate dosage
Time of blood vessel dilation | The measurement of the brachial artery vasodilation time (Cruz 2016; Iida 2006) was made before (baseline), immediately after and every two minutes until completing 20 minutes of evaluation after photobiomodulation
  The duration of the vasodilation of brachial artery after photobiomodulation

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Study Director — Federal University of Health Science of Porto Alegre; Melina Hauck, Me, Principal Investigator — Federal University of Health Science of Porto Alegre; Jociane Schardong, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre; Camila B Bozzetto, Me, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Federal University of Health Science of Porto Alegre (UFCSPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauck M, Schardong J, Donini G, Normann TC, Plentz RDM. Effects of photobiomodulation therapy (PBMT) over endothelial function in healthy individuals: a preliminary crossover clinical trial. Lasers Med Sci. 2023 Apr 19;38(1):104. doi: 10.1007/s10103-023-03762-w. PMID 37072603